CLINICAL TRIAL: NCT02278965
Title: Pilot Biomarker Modulation Study of Metformin and Omega-3 Fatty Acids in Woman With a History of Early Stage Breast Cancer
Brief Title: Metformin and Omega-3 Fatty Acids in Woman With a History of Early Stage Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Katherine D. Crew (Other)
Responsible Party: Sponsor-Investigator, Katherine D. Crew, Assistant Professor of Medicine and Epidemiology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAL2650
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Stage 0 Breast Carcinoma; Breast Neoplasms; Stage I Breast Carcinoma; Stage II Breast Carcinoma; Stage III Breast Carcinoma
Keywords: Breast Cancer; Early Stage
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms | interventions — Metformin; Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Main Arm (Experimental): Open Label- Metformin and Omega-3 fatty acids for 12 months post baseline data collection.
  Interventions: Drug: Metformin; Drug: Omega-3 fatty acids

INTERVENTIONS:
Drug: Metformin — Metformin 850mg, oral, twice a day for 12 months
  Other Names: N,N-dimethyl biguanide hydrochloride
Drug: Omega-3 fatty acids — Omega-3 fatty acids 2 capsules (560 mg each) oral, twice a day for 12 months
  Other Names: Docosahexaenoic acid (DHA)/eicosapentaenoic acid (EPA)

SUMMARY:
The purpose of this study is to determine whether it is feasible to give a combination of Metformin and omega-3 fatty acids for one year to women with a history of early stage breast cancer. We will also evaluate whether the metformin and omega-3 fatty acids combination causes changes in breast tissue, blood, and mammograms.

DETAILED DESCRIPTION:
Metformin is a medication used to treat and prevent diabetes and omega-3 fatty acids has been shown to lower cholesterol and improve cardiovascular health. Research has shown that Metformin and omega-3 fatty acids may also be effective in preventing cancer. In this study, we want to find out what effects, good and/or bad, the Metformin and omega-3 fatty acids combination has on you and your risk of developing a new breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically-confirmed stage 0, I, II, or III breast carcinoma without evidence of disease at trial entry. Participants with a resected local recurrence are eligible
* Minimum of 6 months since last chemotherapy, biologic therapy (i.e., trastuzumab), radiation therapy, and/or breast surgery and no evidence of recurrent disease
* Minimum of 6 months since completion of adjuvant tamoxifen (tamoxifen is known to lower mammographic density119-121). Current use of a third generation aromatase inhibitor [AI] (i.e., anastrozole, letrozole, exemestane) is permitted provided that the participant has been on a stable dose for the past 6 months
* Age 21 to 75 years. Both pre- and postmenopausal women will be included in this study. We will exclude perimenopausal women, defined as menstrual cycle irregularity (variable cycle length that differs from normal by more than 7 days) and an Follicle-Stimulating Hormone (FSH) greater than 20 mili international units
* Negative serum pregnancy testing
* Normal mammogram of the contralateral breast within the past 12 months, defined as no new suspicious calcifications or other abnormal findings warranting a breast biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status less than 2
* Participants must have normal organ and marrow function within 28 days prior to randomization
* Body mass index (BMI) greater than or equal to 25 kilograms per meter squared or baseline fasting glucose of less than 126 milligrams per deciliter
* Participants must have a baseline mammographic density greater than or equal to 25 percent based upon the Breast Imaging Reporting and Data System (BIRADS) density score of 2, 3, or 4. Women with a baseline mammographic density of less than 25 percent (BIRADS Score= 1) will not be eligible
* Willingness to abstain from all omega-3 fish oil supplements for 30 days prior to baseline evaluation and during the study intervention
* Willingness to comply with all study interventions and follow-up procedures
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* History of histologically-confirmed bilateral breast cancer
* History of or plans for bilateral mastectomies
* Evidence of metastatic breast cancer
* Prior radiation therapy or implant in the contralateral breast
* Known diabetes (type 1 or 2) or baseline fasting glucose greater than 126 milligrams per deciliter
* Any condition associated with increased risk of metformin-associated lactic acidosis (e.g., congestive heart failure defined as New York Heart Association [NYHA] Class III or IV functional status, history of acidosis of any type, intake of 3 or more alcoholic beverages per day on average over the past 6 months)
* Currently taking metformin, sulfonylureas, thiazolidinediones, or insulin for any reason
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin or omega-3 fatty acids
* Receiving hormone replacement therapy, tamoxifen, or raloxifene within 6 months of trial entry
* Participants may not be receiving any other investigational agents for 30 days prior to baseline evaluation and during the study intervention
* Any omega-3 fatty acids should not be taken for 30 days prior to baseline evaluation and during the study intervention. If participants are consuming any of these items and would like to participate in this study, then a 30-day washout period will be required. - Uncontrolled or significant co-morbid illness patients receiving active chemotherapy or radiotherapy; or psychiatric illness/social situations that would limit compliance with study requirements

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Number of participants successfully completing the 1-year intervention | 12 months (approximately)
  The primary objective is to assess the safety and feasibility of a one-year intervention of metformin and omega-3 fatty acids in early stage breast cancer patients who completed adjuvant treatment.

SECONDARY OUTCOMES:
Percent in reduction of mammographic density | baseline, 12 months
  Determine the efficacy of these drug interventions in reducing mammographic density
Change in fasting serum insulin microunits per milliliter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating markers of insulin signaling.
Change in C-peptide nanograms per milliliter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating markers of insulin signaling.
Change in insulin-like growth factor 1 (IGF-1) nanograms per milliliter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating markers of insulin signaling.
Change in insulin-like growth factor binding protein 1 (IGFBP-1) nanograms per milliliter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating markers of insulin signaling.
Change in insulin-like growth factor binding protein 3 (IGFBP-3) milligrams per liter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating markers of insulin signaling.
Change in fasting serum glucose milligrams per deciliter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating metabolic profile markers.
Change in total cholesterol milligrams per deciliter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating metabolic profile markers.
Change in high-density lipoprotein (HDL) milligrams per deciliter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating metabolic profile markers.
Change in low-density lipoprotein (LDL) milligrams per deciliter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating metabolic profile markers.
Change in Leptin microunits per liter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating metabolic profile markers.
Change in adiponectin micrograms per milliliter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating metabolic profile markers.
Change in serum C-reactive protein milligrams per deciliter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating inflammatory markers.
Change in Interleukin-6 picograms per milliliter | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating inflammatory markers.
Change in body mass index (BMI) | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating anthropometric measures.
Change in systolic blood pressure | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating anthropometric measures.
Change in diastolic blood pressure | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating anthropometric measures.
Change in homeostatus model assessment (HOMA) score | baseline, month 3, 6, 9, and 12
  Determine the efficacy of these drug interventions in modulating anthropometric measures.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Crew, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- See also: Herbert Irving Comprehensive Cancer Center (HICCC) clinical trials page — http://www.hiccc.columbia.edu/clinical-trials/